CLINICAL TRIAL: NCT06893562
Title: Nine-Year Sustainability After Implementing Measures to Prevent Catheter- Associated Urinary Tract Infections and Bladder Distension in Patients with Hip Fracture
Brief Title: Evaluating Nine-Year Sustainability After Implementing Evidence-Based Practices to Prevent Urinary Tract Infections and Overfilling of the Bladder in Patients with Hip Fracture
Status: Not yet recruiting | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, maria frödin, Professor, Sahlgrenska University Hospital
Other Study IDs: 2025-00397-01
Record Dates: First submitted 2025-03-11; First posted 2025-03-25 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Urinary Catheters; Urinary Retention; Adherence; Documentation Skill; Sustainability of Innovations; Hip Fracture; UTI - Urinary Tract Infection
Keywords: Sustainability of Innovations; Hip fracture; Urinary Retention; Catheter Associated Urinary Tract Infection
MeSH Terms: conditions — Urinary Retention; Hip Fractures; Urinary Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients undergoing hip fracture surgery year nine after the intervention started.
  Interventions: Behavioral: Safe Hands and Safe Bladder intervention

INTERVENTIONS:
Behavioral: Safe Hands and Safe Bladder intervention — Evaluating changes in urinary tract infections and bladder distension nine-year after implementing preventive measures

SUMMARY:
This study focuses on evaluating the long-term sustainability of a urinary catheter care bundle designed to prevent urinary tract infections and bladder distension in patients undergoing surgery for hip fractures. The intervention, which included two key innovations-a urinary catheter certificate and a nurse-driven urinary catheter protocol, was implemented between 2015 and 2020 and successfully reduced urinary tract infections and bladder distension, previously published. However, due to the pandemic, the initiative was paused and had to be reintroduced in 2022. Now, the study aims to assess the effectiveness of these preventive measures 9 years after their initial implementation. The research will analyze changes in the incidence of urinary tract infections, bladder distension, catheterisation methods, and documentation practices in patients aged 65 and older. The findings will help inform healthcare policies and may have broader implications for preventing adverse events in other surgical patient groups

ELIGIBILITY:
Inclusion Criteria:

-Hip fracture surgery at the study site, age 65 years and older and cared for in the ortho-geriatric wards.

Exclusion Criteria:

-No catheterisation during hospital stay

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged 65 years and older undergoing hip fracture surgery at a university hospital in Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Describe changes in the incidence of in-hospital urinary catheter-associated infections; Year 9 will be compared with previously published data from Years 1-5 | For one year
  Definition: Urinary tract infection with onset on day 3 after admission with prior urinary catheterisation. A physician prescribed antimicrobial agents for a urinary tract infection during the hospital stay. Data will be collected from patients' medical records.
  Logistic regression analysis will be performed

SECONDARY OUTCOMES:
Changes in the incidence of in-hospital acquired bladder distension will be compared; Year 9 will be compared to previously published data from Years 1-5. | For one year.
  Definition: Bladder distension is defined according to the national marker for point prevalence measurement when assessing adverse events. Bladderscan volume from patients' medical records.
Changes in urine volume of 500ml and more during hospital stay. Year nine will be compared yera 1-5, previous published data | For one year
  Bladderscan volume from patients' medical records.
Changes in catheterization methods during the hospital stay will be compared, with data from Year 9 compared to previously published data from Years 1-5 | For one year
  Data will be collected from patients' medical records.
Changes in urinary catheter-related documentation in Year 9 will be compared to previously published data from Years 1-5. | For one year
  Catheter-related documentation will be collected from patients' medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Annette Erichsen, Associate Professor, Principal Investigator — Gothenburg University, Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska Academy, Sahlgrenska University hospital/Mölndal, Mölndal, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Erichsen Andersson A, Gillespie BM, Karlsson M, Malchau H, Nellgard B, Wikstrom E, Rogmark C, Tillander J. Reduction of early surgical site and other care related infections in 3553 hip fracture patients: lessons learned from the 5-year Safe Hands project. Antimicrob Resist Infect Control. 2022 Sep 5;11(1):113. doi: 10.1186/s13756-022-01153-4. PMID 36064457
- [Background] Wikstrom E, Dellenborg L, Wallin L, Gillespie BM, Erichsen Andersson A. The Safe Hands Study: Implementing aseptic techniques in the operating room: Facilitating mechanisms for contextual negotiation and collective action. Am J Infect Control. 2019 Mar;47(3):251-257. doi: 10.1016/j.ajic.2018.08.024. Epub 2018 Nov 16. PMID 30449454
- [Background] Erichsen Andersson A, Frodin M, Dellenborg L, Wallin L, Hok J, Gillespie BM, Wikstrom E. Iterative co-creation for improved hand hygiene and aseptic techniques in the operating room: experiences from the safe hands study. BMC Health Serv Res. 2018 Jan 4;18(1):2. doi: 10.1186/s12913-017-2783-1. PMID 29301519
- [Background] Frodin M, Nellgard B, Rogmark C, Gillespie BM, Wikstrom E, Andersson AE. A co-created nurse-driven catheterisation protocol can reduce bladder distension in acute hip fracture patients - results from a longitudinal observational study. BMC Nurs. 2022 Oct 12;21(1):276. doi: 10.1186/s12912-022-01057-z. PMID 36224550
- [Background] Frodin M, Ahlstrom L, Gillespie BM, Rogmark C, Nellgard B, Wikstrom E, Erichsen Andersson A. Effectiveness of implementing a preventive urinary catheter care bundle in hip fracture patients. J Infect Prev. 2022 Mar;23(2):41-48. doi: 10.1177/17571774211060417. Epub 2022 Feb 15. PMID 35340925